CLINICAL TRIAL: NCT03854604
Title: Evaluation of Perfusion Index as an Objective Measure for Postoperative Pain Assessment in Pediatric Patients Undergoing Adenotonsillectomy. An Observational Study.
Brief Title: Perfusion Index as an Objective Measure for Postoperative Pain Assessment in Pediatric Patients.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Assistant Professor of Anesthesia, SICU & pain management. Kasralainy Faculty of medicine, Cairo University
Other Study IDs: N-110-2018
Record Dates: First submitted 2019-02-16; First posted 2019-02-26 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: postoperative pain assessment — evaluation of the efficacy of PI as an objective measure for postoperative pain assessment in pediatric population undergoing adenotonsillectomy.

SUMMARY:
It has been demonstrated that infants and children experience pain in a similar manner to adults, however it used to be undertreated when compared to adult.

Perfusion Index (PI) derived from pulse plethysmography waveform, represents a ratio of pulsatile signal (during arterial inflow) to non-pulsatile signal. PI can represent the peripheral perfusion dynamics due to change of peripheral vasomotor tone. Low PI values suggest peripheral vasoconstriction and high PI values suggest peripheral vasodilation.

The sympathetic nervous system is inherently involved in the pathophysiological responses evoked by painful stimulation.

In the current study, investigators hypothesise that the PI could be a good objective tool for assessment of postoperative pain in children undergoing adenotonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-II
2. Age 3 to 7 years
3. Children undergoing adenotonsillectomy.

Exclusion Criteria:

1. Parents' refusal.
2. Children with behavioral changes
3. Children with physical developmental delay
4. Children on treatment with sedative or anticonvulsant.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 3-7 years, ASA physical status I or II, undergoing Adenotonsillectomy will be included
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Correlation between postoperative (Children's Hospital of Eastern Ontario Scale ) CHEOPS score and postoperative perfusion index. | the time span between arrival to PACU and for at least two hours postoperative

SECONDARY OUTCOMES:
validity of perfusion index to predict postoperative pain and the need of rescue analgesia | he time span between arrival to PACU and for at least two hours postoperative

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Abeer Ahmed, Cairo
  - Kasr Alainy Faculty of Medicine - Cairo university, Cairo
  - Anesthesia department - Faculty of medicine- Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahmed A, Lotfy A, Elkholy J, Abdelhamid B, Ollaek M. Perfusion index as an objective measure of postoperative pain in children undergoing adenotonsillectomy: a cohort study. J Clin Monit Comput. 2022 Jun;36(3):795-801. doi: 10.1007/s10877-021-00710-3. Epub 2021 Apr 23. PMID 33891250